CLINICAL TRIAL: NCT06612125
Title: Comparison of Positive Pressure Ventilation Strategies in Young Children Undergoing Laparoscopic Inguinal Hernia Repair With Laryngeal Mask Airway: A Prospective Randomized Study
Brief Title: Comparing Different Startegies of Positive Pressure Ventilation in Children
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beni-Suef University (Other)
Responsible Party: Principal Investigator, Mariana Soliman, egypt benisuef, Beni-Suef University
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Other
Other Study IDs: FMBSUREC/01092024/Mansour
Record Dates: First submitted 2024-09-21; First posted 2024-09-25 (Actual); Last update posted 2025-01-09 (Actual); Status verified 2025-01

CONDITIONS: Ventilation Therapy; Complications

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- vCV group (Active Comparator): Pediatric patients in the PCV group(n=30) received pressure-controlled ventilation. The initial parameters will be as follows: the peak inspiratory pressure (PIP) will set to provide a tidal volume of 7 ml/kg , respiratory rate will be 16 breaths/min, inspiratory to expiratory ratio was 1:2 with an upper limit of PIP of 20 cm H2O.
  Interventions: Other: volume controlled ventilation
- PCV group (Active Comparator): Pediatric patients in the PCV group(n=30) received pressure-controlled ventilation. The initial parameters will be as follows: the peak inspiratory pressure (PIP) will set to provide a tidal volume of 7 ml/kg , respiratory rate will be 16 breaths/min, inspiratory to expiratory ratio was 1:2 with an upper limit of PIP of 20 cm H2O.
  Interventions: Other: pressure controlled ventilation
- PCV-VG group (Active Comparator): Pediatric patients in the PCV-VG group (n=30)will be conducted with pressure-controlled volume-guaranteed ventilation, target tidal volume will set at 7 mL/kg, with a respiratory rate of 16 breaths/min and a respiratory ratio of 1:2.
  Interventions: Other: pressure controlled volume grantanteed ventilation

INTERVENTIONS:
Other: volume controlled ventilation — Pediatric patients in the VCV group (n= 30) received volume-controlled ventilation, target tidal volume was set at 7 mL/kg, with a respiratory rate of 16 breaths/min and a respiratory ratio of 1:2.
  Arms: vCV group
Other: pressure controlled ventilation — Pediatric patients in the PCV group(n=30) received pressure-controlled ventilation. The initial parameters will be as follows: the peak inspiratory pressure (PIP) will set to provide a tidal volume of 7 ml/kg , respiratory rate will be 16 breaths/min, inspiratory to expiratory ratio was 1:2 with an upper limit of PIP of 20 cm H2O.
  Arms: PCV group
Other: pressure controlled volume grantanteed ventilation — Pediatric patients in the PCV-VG group (n=30)will be conducted with pressure-controlled volume-guaranteed ventilation, target tidal volume will set at 7 mL/kg, with a respiratory rate of 16 breaths/min and a respiratory ratio of 1:2.
  Arms: PCV-VG group

SUMMARY:
The most basic modes of mechanical ventilation are volume-controlled ventilation (VCV) and pressure-controlled ventilation (PCV). VCV guarantees a target volume of ventilation using a constant flow, but may lead to high peak airway pressure (Ppeak) during the gas insufflation . In PCV mode, on the other hand,

DETAILED DESCRIPTION:
The laryngeal mask airway (LMA) provides a useful alternative for airway management during general anaesthesia. Inflation of the LMA cuff produces a low-pressure seal around the larynx, enabling positive pressure ventilation (PPV). The use of LMA as an airway management technique is common in the pediatric anesthesia because of its less irritating effect on the airways due to its location in the upper larynx. Now, the use of laryngeal mask instead of tracheal intubation for airway management has been achieved in day surgery, therefore, how to perform a respiratory management with a laryngeal mask is particularly important. In addition, mechanical ventilation is also a commonly used method of airway management in clinical practice. the ventilator will deliver a constant pressure by decelerating the flow. However, the ventilation volume varies according to the patient's respiratory mechanics . Pressure-controlled ventilation-volume guaranteed (PCV-VG) combines the advantages of both VCV and PCV, which delivers a stable ventilation volume using a decelerating flow pattern.

ELIGIBILITY:
Inclusion Criteria:

1. age between 1 and 5 years.
2. patient scheduled for laparoscopic inguinal hernia repair.
3. American Society of Anesthesiologists classification of physical status of I-II.

Exclusion Criteria:

1. cardiopulmonary disease.
2. severe hepatorenal dysfunction.
3. history of upper respiratory tract infection 2 weeks before the operation.
4. overweight [more than 20% of standard body weight].
5. neuromuscular disease.
6. anticipated difficult airway.
7. hiatus hernia or gastroesophageal reflux disease.

Ages: 1 Year to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 78 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-03-01 (Estimated); Study Completion 2025-03-30 (Estimated)

PRIMARY OUTCOMES:
(PIP) | within one hour
  peak inspiratory pressure
Pplat | within one hour
  plateau airway pressure
(Cdyn) | within one hour
  pulmonary dynamic compliance
(RAW | within one hour
  airway resistance
VT | within one hour
  exhaled tidal volume
EtCO2 | within one hour
  end-expiratory carbon dioxide
Vd/VT | within one hour
  physiologic dead space over tidal volume

SECONDARY OUTCOMES:
(MAP) | within one hour
  mean arterial pressure
(HR) | within one hour
  heart rate
postoperative respiratory adverse events | within 24 hour
  cough, hoarseness, sore throat, hypoxemia, laryngospasm, bronchospasm.

CONTACTS AND LOCATIONS:
Overall Officials: Mariana as Mansour, MD, Principal Investigator — benisuef university hospital Egypt
Locations (1):
- Benisuef university hospital, Benisuef, Egypt